CLINICAL TRIAL: NCT04322513
Title: Biomarkers Identification for Diagnosis and Treatment of SARS-COV-2 Infection
Brief Title: Biomarkers for Identification of COVID-19 Infection
Acronym: B-DT-COV2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: Azienda Ospedaliera Pugliese Ciaccio (Other); Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, Clinical Professor, University of Catanzaro
Other Study IDs: covid-19 biomarkers
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 positive patients: all drugs used for standard treatment
  Interventions: Diagnostic Test: Biomarkers expression
- Covid-19 negative patients
  Interventions: Diagnostic Test: Biomarkers expression

INTERVENTIONS:
Diagnostic Test: Biomarkers expression — Evaluation in biomarkers expression between 2 groups

SUMMARY:
Acute lung injury represents the most severe form of the viral infection sustained by coronavirus disease 2019 (Covid-19) also named as SARS-CoV-2, a new virus emerged in December 2019 in Wuhan (China). The diagnosis is clinical and patients develop flu-like syndrome with fever and cough; patients with clinical symptoms can perform a swab test, including molecular and/or antigen swab, for diagnosis of positivity to Covid-19. Even if diagnosis and treatment are well described, to date, this viral pandemic infection induces an increased mortality in the world. The aim of the present project is to evaluate specific biomarkers that could be used for patient stratification and for tailor therapy in COVID-19 infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years, extremes included, male or female In conscious patients, ability to understand and the willingness to sign a written informed consent document; in unconscious patients informed consent will be signed from parents or legal tutors.

Exclusion Criteria:

* Patients that don't sign the informed consent

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both sexes and > 18 years with and without covid-19 infection that came in hospital for flu-like syptoms: cough fever and dyspnea
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Biomarkers expression | up to 30 days
  Change in biomarkers (microRNAs, oxidative stress, Neuron-Specific Enolase, IL-2, IL-6, TNF-alfa, leukocytes, subtypes lymphocytes) in covid-19 positive patients vs covid-negative patients
Liver Biomarkers expression | up to 30 days
  Change in CYP450 expression in covid-19 positive patients that develop adverse drug reactions or drug inefficacy

SECONDARY OUTCOMES:
biomarkers expression (microRNAs, oxidative stress, Neuron-Specific Enolase, IL-2, IL-6, TNF-alfa, leukocytes, subtypes lymphocytes) after treatment | 60 days
  Changes in biomarkers in covid-19 patients before and after standard treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Luca Gallelli, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No